CLINICAL TRIAL: NCT07059364
Title: Empowering Caregivers to Promote Child Independence and Persistence With Activities
Brief Title: Empowering Caregivers to Promote Child Independence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Autism Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0708-24-FB; PRO-25-006 (Other Grant/Funding Number: Autism Science Foundation)
Record Dates: First submitted 2025-06-09; First posted 2025-07-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-07

CONDITIONS: Profound Autism
Keywords: Profound Autism; Picture-Based Activity Schedules; Caregiver Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to caregiver activity schedules training (CAST) or treatment as usual (TAU) in a 1:1 ratio according to permuted blocks. CAST consists of 40 hours of intervention in 2-hour appointments, 3-5 days/week, for 3-6 weeks. The appointment frequency and duration are intended to provide caregivers with flexibility and promote access to research. The TAU group will be offered CAST after their final assessment visit.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as Usual (TAU) will consist of 3-6 weeks of continuing usual care.
- Caregiver Activity Schedules Treatment (Experimental): Caregiver Activity Schedules Treatment (CAST) consists of a picture-based activity schedule compiled into binders created for each participant. Activities for each participant will be selected with caregivers to include preference and feasibility. Activity steps include 1) opening the schedule/turning the page, 2) orienting to the picture, 3) retrieving the activity, 4) completing the activity, 5) putting the activity away, and 6) repeating each step until all activities are completed. Graduated guidance without verbal prompts will be used to support schedule completion. Implementer proximity will be faded within and between sessions. Caregivers will receive written descriptions of procedures. The researcher will describe and model all procedures and answer questions. Caregivers will implement procedures with their child and receive in-vivo feedback.
  Interventions: Behavioral: CAST Treatment

INTERVENTIONS:
Behavioral: CAST Treatment — Activity completion will be evaluated based the number of consecutive and total activities completed, duration of sustained activity engagement, prompts or redirection, and adult proximity at baseline and post-trial.
  Arms: Caregiver Activity Schedules Treatment

SUMMARY:
The proposed study aims to address the unique needs of caregivers and their adolescent children with profound autism. The constant supervision and 24/7 care that caregivers need to provide their children to ensure their health and safety often leaves little time for household duties, self-care routines, and spending time with family and friends. Investigators aim to alleviate the vigilant monitoring provided by caregivers for brief periods by increasing their child's independent, sustained engagement in meaningful activities and improving the quality of life for both adolescents with profound autism and their caregivers. Caregivers will either receive training to use picture-based activity schedules or continue with their usual routines. After the study, caregivers who continued their usual routines will also be offered the training. Investigators will evaluate the feasibility and acceptability of the training based on the children's performance, pre- and post-study improvement ratings, and caregiver feedback.

DETAILED DESCRIPTION:
Approximately 25% of children with autism are estimated to meet the criteria for profound autism. Profound autism describes those with the greatest support needs because of the coinciding significant intellectual disability and limited/absent verbal communication. Because individuals with profound autism have been excluded from research, the investigator's understanding of effective assessments and interventions for this population and their families is incomplete. One defining feature associated with caring for a child with profound autism is the 24/7 supervision required from caregivers, often described as a feeling of constant vigilance. Although previous research on the matter may not use the specific term, profound autism, much can be gleaned from studies of caregivers with adult autistic children who cannot be left alone, autistic children with co-occurring intellectual disability, or older studies including children with IQ scores below 50 before autism was well understood. Caregivers facing these 24/7 obligations experience increased time constraints that prevent their self-care routines, limit time with family and friends, and reduce time spent on personal interests and work-related activities. Caregivers also report reduced time spent sleeping, preparing meals, and completing other household duties. Some report being unable to leave their child unattended for as little as 5 minutes. Relatedly, caregivers of profoundly autistic children report some of their greatest hopes for their children to be increased independence and autonomy to engage in enjoyable activities. Teaching autistic children how to engage appropriately with items can increase independent leisure engagement and increasing sustained activity engagement can promote autonomy and overall well-being. Therefore, interventions that promote independent, sustained engagement with activities could simultaneously benefit people with profound autism and their caregivers. However, characteristic restricted interests and repetitive behaviors can impede sustained activity engagement and interfere with transitioning to new activities. Thus, additional environmental supports, such as visuals, are sometimes needed. Picture-based activity schedules are an evidence-based practice that promotes sustained engagement with activities with reduced adult assistance. However, additional research is necessary to evaluate this intervention for individuals with profound autism and their caregivers.

The proposed study focuses on alleviating vigilant-level supervision provided by caregivers for brief periods while simultaneously increasing independent, sustained engagement with meaningful activities for their adolescent children with profound autism. Participants will randomly be assigned to either the Caregiver Activity Schedules Treatment (CAST) group and receive 40 hours of training in picture-based activities or be assigned to the Treatment as Usual (TAU) group. The TAU group will be offered CAST training following the trial. The feasibility, acceptability, and preliminary efficacy will be evaluated using measures of participant performance, participant affect, clinician ratings, and independent evaluation by an expert using the Clinical Global Impressions Improvement Scale (CGI-I).

ELIGIBILITY:
Inclusion Criteria:

* Autistic individuals 10 to 17 years of age
* Severe or profound intellectual disability diagnosis or reportedly in line with diagnostic criteria based on Autism Diagnostic Observation Schedule, Second Edition ADOS-2
* Developmental Profile 4 (DP-4) Cognitive/Communication Domain scores below 70 (Delayed)
* Adaptive Behavior Assessment System (ABAS-3) Communication, Health and Safety, and Leisure Domains adaptive skill scores in the Low to Extremely Low range
* Can complete between 3-10 simple leisure or daily living skill tasks or activities independently (caregiver may prompt or provide oversight)
* Caregivers can remain present to assist with toileting if more than one person is needed to assist
* No medication or stable medication regimen with no planned changes for study duration
* Stable intervention and/or educational services with no planned changes for study duration
* English spoken by at least one caregiver

Exclusion Criteria:

* Known serious medical condition or serious behavioral/psychiatric condition requiring immediate alternative focused intervention

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participant Accrued | Until accrual is complete, approximately 1 year
  Number of caregivers who accept random assignment as determined by refusal rate of eligible participants.
Rate of Participant Attrition | Up to 6 weeks
  Participant attrition rate will be determined over the course of the study.
Ratings of Caregiver Activity Schedules Treatment Acceptability | Up to 6 weeks
  The acceptability of the Caregiver Activity Schedules Treatment (CAST) intervention by the caregiver will be measured using a 1 to 5 scale (anchored by 1 strongly disagree, and 5, strongly agree) by average ratings of agree (4) or strongly agree (5) to all acceptability rating scale statements and adolescents willingness to participate in intervention sessions.
Caregiver Reported Continued Use of Activity Schedules Treatment | Up to 6 weeks
  The reported continued use of the Caregiver Activity Schedules Treatment activity schedules at home by the caregiver will be determined at 6-weeks by responses to a 5 question open-ended questionaire.

SECONDARY OUTCOMES:
Total Number of Activities Completed | Baseline (enrollment) to end of treatment, up to 6 weeks
  Caregiver Activity Schedules Treatment (CAST) activity completion will be evaluated based the number of total activities completed at baseline and post-trial.
Number of Consecutive Activities Completed | Baseline (enrollment) to end of treatment, up to 6 weeks
  Caregiver Activity Schedules Treatment (CAST) activity completion will be evaluated based the number of consecutive activities completed at baseline and post-trial.
Duration of Sustained Activity Engagement | Baseline (enrollment) to end of treatment, up to 6 weeks
  Caregiver Activity Schedules Treatment (CAST) activity completion will be evaluated based the duration of sustained activity engagement at baseline and post-trial.
Number of Prompts to Complete Activities | Baseline (enrollment) to end of treatment, up to 6 weeks
  Caregiver Activity Schedules Treatment (CAST) activity completion will be evaluated based the number of prompts needed to complete activities at baseline and post-trial.
Number of Redirections to Stay on Task | Baseline (enrollment) to end of treatment, up to 6 weeks
  Caregiver Activity Schedules Treatment (CAST) activity completion will be evaluated based the number of redirections to stay on task at baseline and post-trial.
Caregiver Proximity to Their Child | Baseline (enrollment) to end of treatment, up to 6 weeks
  Caregiver Activity Schedules Treatment (CAST) activity completion will be evaluated based the caregiver proximity to their child at baseline and post-trial.
Improvement Ratings on the Clinical Global Impressions - Improvement Scale | Baseline (enrollment) to end of treatment, up to 6 weeks
  The Clinical Global Impressions - Improvement Scale (CGI-I) is a 7-point scale designed to measure overall improvement from baseline. Scores range from 1 (Very Much Improved) to 7 (Very Much Worse). An independent evaluator (IE) will assess data recorded from direct observation (i.e., number of activities completed, duration of sustained engagement, amount and type of adult support provided) of the participant and caregiver at baseline and post-trial. Additionally, the IE will consider the baseline and post-trial Parent Target Problems (PTP) narratives which document caregiver-nominated target problems in specific areas of concern identified through conversation with caregivers. Using this information from baseline and post trial, the IE will yeild an improvement rating on the CGI-I.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Shillingsburg, PhD, BCBA-D, Principal Investigator — University of Nebraska
Locations (1):
- Munroe-Meyer Insitute University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
All study outcome measures will be shared with the National Database for Autism Reserch. Global Unique Identifiers will be used to share data from the study and all indentifying participant information will be removed before sharing.
Time Frame: October 1, 2025
Access Criteria: All IPD and supporting information will be availabile in the open science data repository the National Database for Autism Research (NDAR)
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Scahill L, Shillingsburg MA, Ousley O, Pileggi ML, Kilbourne RL, Buckley D, Gillespie SE, McCracken C. A Randomized Trial of Direct Instruction Language for Learning in Children With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2022 Jun;61(6):772-781. doi: 10.1016/j.jaac.2021.11.034. Epub 2022 Jan 31. PMID 35093490
- [Background] Bearss K, Johnson C, Smith T, Lecavalier L, Swiezy N, Aman M, McAdam DB, Butter E, Stillitano C, Minshawi N, Sukhodolsky DG, Mruzek DW, Turner K, Neal T, Hallett V, Mulick JA, Green B, Handen B, Deng Y, Dziura J, Scahill L. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. JAMA. 2015 Apr 21;313(15):1524-33. doi: 10.1001/jama.2015.3150. PMID 25898050
- [Background] Sheridan E, Gillespie S, Johnson CR, Lecavalier L, Smith T, Swiezy N, Turner K, Pritchett J, Mruzek DW, Evans AN, Bearss K, Scahill L. Using Parent Target Problem Narratives to Evaluate Outcomes in Children with Autism Spectrum Disorder. Res Child Adolesc Psychopathol. 2021 Nov;49(11):1527-1535. doi: 10.1007/s10802-021-00843-8. Epub 2021 Jul 2. PMID 34213717
- [Background] Hirst K, Zamzow RM, Stichter JP, Beversdorf DQ. A Pilot Feasibility Study Assessing the Combined Effects of Early Behavioral Intervention and Propranolol on Autism Spectrum Disorder (ASD). Children (Basel). 2023 Sep 30;10(10):1639. doi: 10.3390/children10101639. PMID 37892301
- [Background] Shillingsburg MA, Hansen B, Wright M. Rapport Building and Instructional Fading Prior to Discrete Trial Instruction: Moving From Child-Led Play to Intensive Teaching. Behav Modif. 2019 Mar;43(2):288-306. doi: 10.1177/0145445517751436. Epub 2018 Jan 17. PMID 29338313
- [Background] Gordon KR, Shillingsburg MA. Teaching mands for social information to individuals with develop mental disabilities. Adv Neurodev Disord. 2019;3;363-371. doi: 10.1007/s41252-019-00126-w
- [Background] Frampton SE, Shillingsburg MA, Simeone PJ. Feasibility and Preliminary Efficacy of Direct Instruction for Individuals With Autism Utilizing Speech-Generating Devices. Behav Anal Pract. 2020 Feb 11;13(3):648-658. doi: 10.1007/s40617-020-00412-3. eCollection 2020 Sep. PMID 32953393
- [Background] Shillingsburg MA, Frampton SE, Juban B, Weddle SA, Silva MR. Implementing an applied verbal behavior model in classrooms. Behav Intervent. 2022;37(1), 56-78. doi.org/10.1002/bin.1807
- [Background] Koyama T, Wang HT. Use of activity schedule to promote independent performance of individuals with autism and other intellectual disabilities: a review. Res Dev Disabil. 2011 Nov-Dec;32(6):2235-42. doi: 10.1016/j.ridd.2011.05.003. Epub 2011 Jun 6. PMID 21645988
- [Background] Lequia J, Machalicek W, Rispoli MJ. Effects of activity schedules on challenging behavior exhibited in children with autism spectrum disorders: A systematic review. Res Autism Spectr Disord. 2012;6(1); 480- 492. doi: 10.1016/j.rasd.2011.07.008
- [Background] . Cho S, Noor NHBM, Sonoyama S. A review of activity schedules for individuals with autism spectrum disorder. J of Spec Educ Resear. 2017;5(2):65-76. doi:10.6033/specialeducation.5.65
- [Background] Cavalari RN, Romanczyk RG. Caregiver perspectives on unintentional injury risk in children with an autism spectrum disorder. J Pediatr Nurs. 2012 Dec;27(6):632-41. doi: 10.1016/j.pedn.2011.07.013. Epub 2011 Sep 13. PMID 23101727
- [Background] Knight V, Sartini E, Spriggs AD. Evaluating visual activity schedules as evidence-based practice for individuals with autism spectrum disorders. J Autism Dev Disord. 2015 Jan;45(1):157-78. doi: 10.1007/s10803-014-2201-z. PMID 25081593
- [Background] Lang R., O'Reilly M, Rispoli M, Shogren K., Machalicek W, Sigafoos J, Regester A. Review of interventions to increase functional and symbolic play in children with autism. Educ and Train in Dev Disab. 2009;44;481-492. https://www.jstor.org/stable/24234257
- [Background] Schwartz IS, Kelly EM. Quality of life for people with disabilities: Why applied behavior analysts should consider this a primary dependent variable. Resear and Pract Severe Disabil. 2021;46(3);159-172. doi.org/10.1177/15407969211033629
- [Background] Edwards CK, Landa RK, Frampton SE, Shillingsburg MA. Increasing Functional Leisure Engagement for Children With Autism Using Backward Chaining. Behav Modif. 2018 Jan;42(1):9-33. doi: 10.1177/0145445517699929. Epub 2017 May 3. PMID 28466648
- [Background] Celia T, Freysteinson W, Fredland N, Bowyer P. Battle weary/battle ready: A phenomenological study of parents' lived experiences caring for children with autism and their safety concerns. J Adv Nurs. 2020 Jan;76(1):221-233. doi: 10.1111/jan.14213. Epub 2019 Oct 27. PMID 31566790
- [Background] Vaz S, Thomson A, Cuomo B, Falkmer T, Chamberlain A, Black MH. Co-occurring intellectual disability and autism: Associations with stress, coping, time use, and quality of life in caregivers. Research in ASD. 2021; 84;101765. doi.org/10.1016/j.rasd.2021.101765
- [Background] Marsack-Topolewski CN, Church HL. Impact of Caregiver Burden on Quality of Life for Parents of Adult Children With Autism Spectrum Disorder. Am J Intellect Dev Disabil. 2019 Mar;124(2):145-156. doi: 10.1352/1944-7558-124.2.145. PMID 30835531
- [Background] Dupont A. A study concerning the time-related and other burdens when severely handicapped children are reared at home. Acta Psychiatrica Scandinavia. 1980;62(Suppl. 285);249-257.
- [Background] Dudley, Carolyn and Emery, J. C. Herbert.The Value of Caregiver Time: Costs of Support and Care for Individuals Living with Autism Spectrum Disorder. SPP Research Paper. 2014; 7-1. doi.org/10.2139/ssrn.2379633
- [Background] Lord C, Charman T, Havdahl A, Carbone P, Anagnostou E, Boyd B, Carr T, de Vries PJ, Dissanayake C, Divan G, Freitag CM, Gotelli MM, Kasari C, Knapp M, Mundy P, Plank A, Scahill L, Servili C, Shattuck P, Simonoff E, Singer AT, Slonims V, Wang PP, Ysrraelit MC, Jellett R, Pickles A, Cusack J, Howlin P, Szatmari P, Holbrook A, Toolan C, McCauley JB. The Lancet Commission on the future of care and clinical research in autism. Lancet. 2022 Jan 15;399(10321):271-334. doi: 10.1016/S0140-6736(21)01541-5. Epub 2021 Dec 6. No abstract available. PMID 34883054
- [Background] Hughes MM, Shaw KA, DiRienzo M, Durkin MS, Esler A, Hall-Lande J, Wiggins L, Zahorodny W, Singer A, Maenner MJ. The Prevalence and Characteristics of Children With Profound Autism, 15 Sites, United States, 2000-2016. Public Health Rep. 2023 Nov-Dec;138(6):971-980. doi: 10.1177/00333549231163551. Epub 2023 Apr 19. PMID 37074176